CLINICAL TRIAL: NCT01637168
Title: Clinical Phase III, Randomized, Double-blind, Prospective Study, for Efficacy and Safety Evaluation of Panax Ginseng + Associations Compared to Ginkgo Biloba in Symptomatic Cognitive Function Disorder Treatment.
Brief Title: Comparison of the Panax Ginseng + Associations to Ginkgo Biloba in the Treatment of Cognitive Function Disorders
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Canceled [By sponsor decision)
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GGKEMS0910
Record Dates: First submitted 2012-03-29; First posted 2012-07-11 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Memory Deficit
Keywords: Disorders of cognitive function
MeSH Terms: conditions — Memory Disorders | interventions — Asian ginseng; Ginkgo Extract; Geritol; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group (Experimental): Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamin - 1 tablet, 2 times a day (12/12 hours).
  Interventions: Drug: Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamin
- Comparator Group (Active Comparator): Ginkgo Biloba (Tebonin ®) - 1 tablet, 2 times a day (12/12 hours).
  Interventions: Drug: Ginkgo Biloba (Tebonin®)

INTERVENTIONS:
Drug: Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamin — A tablet, 2 times daily (12/12 hours).
  Arms: Test Group
Drug: Ginkgo Biloba (Tebonin®) — A tablet, 2 times daily (12/12 hours).
  Other Names: Ginkgo Biloba
  Arms: Comparator Group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two different drugs in the treatment of patients diagnosed with memory difficulties and a decline in cognitive function.

This is a parallel distribution: a group of patients will be treated with a combination Panax Ginseng + Ginkgo Biloba + multivitamin + Polyminerals (EMS), and another group with Ginkgo Biloba (Tebonin ®).

DETAILED DESCRIPTION:
STUDY DESIGN:

* multicenter, phase III, double-blind, randomized entry of patients, prospective and comparative
* The duration of the study: 60 days
* 3 visits (days 1, 30 and 60)
* Evaluate the effectiveness of the association
* Evaluate the safety of the combination
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any race, sex, aged 18-60 years;
2. Patients presenting two or more symptoms associated with disorders of cognitive function such as memory impairment, poor concentration, depressed mood, decreased mental capacity, provided they score value is below 24 in the evaluation of the psychometric test (Mini Test-mental and WMS-R Logical Memory);
3. Consent of the patient (Signature of the IC);
4. Patients are able to read and write;
5. "Washout" of at least two weeks of the start of the study, in case of use of multivitamins or any other medication for symptomatic treatment of disorders of cognitive function.
6. Women of childbearing potential must submit βHCG negative serum;
7. Patients are able to understand and carry out the study procedures;

Exclusion Criteria:

1. Patients with hypersensitivity to the components of the formula;
2. Patients who are making use of levodopa or salicylates;
3. Routine use of medications that alter cognitive functions such as barbiturates, anticonvulsants, benzodiazepines, neuroleptics, alcohol and illicit drugs;
4. Pregnant or lactating women;
5. Participation in another clinical trial with investigational medication in the last 3 months;
6. Patients with prior knowledge of infectious disease;
7. Patients who are taking other multivitamins or any other medications for the symptomatic treatment of disorders of cognitive function, at least two weeks prior to study initiation.
8. Patients with organic dementias such as Alzheimer's, Pick's disease, Creutzfeldt-Jacob Disease, Huntington's, Parkinson's disease, dementia caused by human immunodeficiency virus (HIV), hypothyroidism, vascular dementia (arteriosclerotic dementia), dementia senile among others;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Study to evaluate the efficacy and safety of the association Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamins compared to Ginkgo Biloba (Tebonin ®) for the symptomatic treatment of disorders of cognitive function. | 60 days
  To evaluate the efficacy of the association between Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamin to treat patients with disorders of cognitive function compared to treatment with the drug Ginkgo Biloba (Tebonin ®)
  The assessment of effectiveness will be determined by statistical evaluation of the scores of responses related to quality of life questionnaires and psychometric tests (Mini-Mental Test and Test of Logical Memory WMS-R).

SECONDARY OUTCOMES:
Study to evaluate the efficacy and safety of the association Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamins compared to Ginkgo Biloba (Tebonin ®) for the symptomatic treatment of disorders of cognitive function. | 60 days
  To evaluate the safety of the association between Panax Ginseng + Ginkgo Biloba + Polyminerals + Multivitamin to treat patients with disorders of cognitive function compared to treatment with the drug Ginkgo Biloba (Tebonin ®).
  The safety of the medication to be prescribed by the observation of adverse events and related to the study medication. Analysis of safety tests (biochemical profile, complete blood count, blood glucose, cholesterol and uric acid) requested at visit 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Felício MD Savioli Neto, Principal Investigator — Clínica Dr. Felício Savioli
Locations (1):
- Cliníca Dr. Felício Savioli, Cotia, São Paulo, Brazil